CLINICAL TRIAL: NCT06241534
Title: Evaluation of the Effectiveness of Modern Technologies in Psychologically-enhanced Rehabilitation in Patients With Cardiovascular Diseases
Brief Title: Supporting Methods in Cardiovascular Diseases Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Gajda-Med District Hospital (Unknown); Cardiology Center Pro Corde (Unknown); Healthcare Innovation Technology Lab, IRCCS San Camillo Hospital (Unknown)
Responsible Party: Principal Investigator, Adam Wrzeciono, MSc, MSc, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT/CR/01/2023
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Mood Disorders; Depressive Symptoms; Anxiety; Stress
Keywords: cardiac rehabilitation; psychotherapy; therapeutic recordings; virtual reality; depression; anxiety; stress
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Mood Disorders; Depression; Anxiety Disorders | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recordings Group (Experimental): Cardiac rehabilitation supplemented by relaxation-therapeutic recordings
  Interventions: Behavioral: Cardiac rehabilitation; Behavioral: Relaxation-therapeutic recordings
- VR Group (Experimental): Cardiac rehabilitation supplemented by VR therapy
  Interventions: Behavioral: Cardiac rehabilitation; Device: Virtual reality therapy
- Control Group (Active Comparator): Cardiac rehabilitation supplemented by Schultz Autogenic Training
  Interventions: Behavioral: Cardiac rehabilitation; Behavioral: Schultz Autogenic Training

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Four weeks of cardiac rehabilitation conducted in an outpatient care facility. Three times per week (80 minutes per day) cardiologically monitored aerobic training consisting of: 40 minutes of interval training on a cycloergometer and 40 minutes of general fitness exercises.
Behavioral: Relaxation-therapeutic recordings — 8 sessions of relaxation-therapeutic recordings in the non-sleep deep rest concept.
  The content of the recording is based on the 'body scanning technique', which constitutes the core of the therapy. This approach aims to quiet the overactive sympathetic part of the autonomic nervous system. During therapy, the patients take a 'journey' through their own body from feet to head. Following the voice of the narrator, the patient focuses on specific body parts, tries to feel this place and then relaxes tense muscles. Relaxation of individual body parts (muscle groups) is combined with breathing exercises. Conscious and mindful breathing deepens the state of relaxation. Additionally, the recording includes therapeutic suggestions related to making a choice between: overload and relief, holding on and letting go, acting and sensing. Furthermore, suggestions focus the patient on inner wisdom that allows them to make the best decisions.
  Arms: Recordings Group
Device: Virtual reality therapy — 8 sessions of VR therapy (each of them 20 minutes long). As a virtual reality source, VR TierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach.The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
  Arms: VR Group
Behavioral: Schultz Autogenic Training — 8 sessions of Schultz Autogenic Training (each of them 20 minutes long).
  Arms: Control Group

SUMMARY:
The study evaluates how various therapeutic approaches perform in addressing depression, anxiety symptoms, and stress levels among patients in the second stage of cardiac rehabilitation. This study aims to evaluate the influence of the used therapeutic approaches on psychological outcomes and to compare the effectiveness of these therapies.

DETAILED DESCRIPTION:
Depression, anxiety, and high levels of perceived stress are increasingly common problems associated with cardiovascular disease (CVD). The relationship between anxiety-depressive disorders and the risk of CVD is confirmed by behavioral and physiological mechanisms. According to the American Heart Association, depression is a negative prognostic factor at all stages of treatment of CVD. The most important risks in people with CVD and anxiety-depressive disorders, as comorbidities, are an increased risk of recurrent cardiovascular events and increased mortality. However, psychological disorders in patients with CVD are still not sufficiently diagnosed and, consequently, are not adequately treated. Therefore, it is necessary to look for effective methods to support cardiac rehabilitation from a psychological perspective.

The first group of patients will receive relaxation-therapeutic recordings (referred to as the Recording Group) in addition to monitored cardiac physical training. The second group will receive virtual reality (VR) therapy (referred to as the VR Group) alongside monitored cardiac physical training. The third group (referred to as the Control Group) will receive Schultz Autogenic Training as a standard supplement to cardiological training.

The aims of the study:

1. The evaluation of the influence of relaxation-therapeutic recordings on the anxiety-depressive symptoms and the stress level of the patients undergoing second stage of cardiac rehabilitation.
2. The comparison of the effectiveness of therapeutic recordings with the effectiveness of VR therapy and Schultz Autogenic Training.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Disease;
* the second stage of cardiac rehabilitation conducted in outpatient settings

Exclusion Criteria:

* inability to self-complete the research questionnaires;
* presence of the following issues at the time of the examination or in the medical data: disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders;
* initiation of psychiatric treatment during the research project;
* contraindications for virtual therapy (epilepsy, vertigo, eyesight impairment);
* the patient's refusal at any stage of the research project.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale Hospital Anxiety and Depression Scale | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.
Perception of Stress Questionnaire | 20 minutes
  The Perception of Stress Questionnaire (PSQ) was created by Plopa and Makarowski. It is a 27-item scale scoring from 1 to 5 points for each item, where 21 items examine the level of stress in the areas of emotional tension, external stress and intrapsychic stress, and six items refer to the lie scale. The global scoring for the perception of stress ranges from 21 to 105, with a cut-off point of 60 for an elevated level of perceived stress. Higher scores indicate higher stress perception.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Prof., Study Director — Wroclaw University of Health and Sport Sciences; Adam Wrzeciono, MSc., Principal Investigator — Wroclaw University of Health and Sport Sciences; Sandra Jóźwik, Ph.D., Principal Investigator — Cardiology Center Pro Corde; Błażej Cieślik, Ph.D., Study Chair — Healthcare Innovation Technology Lab, IRCCS San Camillo Hospital; Paweł Kiper, Ph.D., Study Chair — Healthcare Innovation Technology Lab, IRCCS San Camillo Hospital; Robert Gajda, Prof., Study Director — Gajda-Med District Hospital
Locations (1):
- Cardiology Center Pro Corde, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Natt Och Dag Y, Mehlig K, Rosengren A, Lissner L, Rosvall M. Negative emotional states and negative life events: Consequences for cardiovascular health in a general population. J Psychosom Res. 2020 Feb;129:109888. doi: 10.1016/j.jpsychores.2019.109888. Epub 2019 Nov 29. PMID 31835155
- [Background] Silverman AL, Herzog AA, Silverman DI. Hearts and Minds: Stress, Anxiety, and Depression: Unsung Risk Factors for Cardiovascular Disease. Cardiol Rev. 2019 Jul/Aug;27(4):202-207. doi: 10.1097/CRD.0000000000000228. PMID 30130257
- [Background] Szczepanska-Gieracha J, Morka J, Kowalska J, Kustrzycki W, Rymaszewska J. The role of depressive and anxiety symptoms in the evaluation of cardiac rehabilitation efficacy after coronary artery bypass grafting surgery. Eur J Cardiothorac Surg. 2012 Nov;42(5):e108-14. doi: 10.1093/ejcts/ezs463. Epub 2012 Aug 19. PMID 22906598
- [Background] Szczepanska-Gieracha J, Jozwik S, Cieslik B, Mazurek J, Gajda R. Immersive Virtual Reality Therapy as a Support for Cardiac Rehabilitation: A Pilot Randomized-Controlled Trial. Cyberpsychol Behav Soc Netw. 2021 Aug;24(8):543-549. doi: 10.1089/cyber.2020.0297. Epub 2021 Feb 11. PMID 33577375
- [Background] Jozwik S, Cieslik B, Gajda R, Szczepanska-Gieracha J. Evaluation of the Impact of Virtual Reality-Enhanced Cardiac Rehabilitation on Depressive and Anxiety Symptoms in Patients with Coronary Artery Disease: A Randomised Controlled Trial. J Clin Med. 2021 May 16;10(10):2148. doi: 10.3390/jcm10102148. PMID 34065625
- [Background] Jozwik S, Cieslik B, Gajda R, Szczepanska-Gieracha J. The Use of Virtual Therapy in Cardiac Rehabilitation of Female Patients with Heart Disease. Medicina (Kaunas). 2021 Jul 28;57(8):768. doi: 10.3390/medicina57080768. PMID 34440974
- [Background] Jozwik S, Wrzeciono A, Cieslik B, Kiper P, Szczepanska-Gieracha J, Gajda R. The Use of Virtual Therapy in Cardiac Rehabilitation of Male Patients with Coronary Heart Disease: A Randomized Pilot Study. Healthcare (Basel). 2022 Apr 16;10(4):745. doi: 10.3390/healthcare10040745. PMID 35455922